CLINICAL TRIAL: NCT03833713
Title: Utilizing Text Messaging to Improve Vehicle Safety Among At-Risk Young Adults
Acronym: SaVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Maria Pacella, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY20020035 (CC); 693JJ91850017 (Other Grant/Funding Number: NHTSA)
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Risk Reduction
Keywords: text message; behavioral intervention; motor vehicle
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, 2-arm (intervention vs. control)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS Intervention (Experimental): Once-weekly automated SMS dialogue sessions or micro-interventions and use behavior change techniques including self-monitoring with performance feedback and goal support
  Interventions: Behavioral: SMS Dialogue
- SMS Assessments (Active Comparator): Once-weekly SMS assessments related to their target risk behavior without receiving any feedback or goal support
  Interventions: Behavioral: SMS Assessments

INTERVENTIONS:
Behavioral: SMS Dialogue — Once-weekly SMS dialogue sessions or micro-interventions and use behavior change techniques (BCTs) including self-monitoring with performance feedback and goal support
  Arms: SMS Intervention
Behavioral: SMS Assessments — Once-weekly SMS assessments of motor vehicle risks
  Arms: SMS Assessments

SUMMARY:
The "Safe Vehicle Engagement (SaVE)" trials are 3 parallel randomized clinical trials that aim to determine the impact of text messaging (SMS) vehicle safety interventions vs. weekly SMS vehicle safety self-monitoring alone on seat belt use, distracted driving and drink driving among young adults identified in the emergency department (ED) with risky vehicle behaviors.

DETAILED DESCRIPTION:
The investigators propose to conduct 3 related randomized, controlled, parallel group, assessor-blind, superiority trials of 6-week text message interventions vs. SMS vehicle safety self-monitoring in young adult participants with risky vehicle behaviors. A total of 500 adult participants will be enrolled: 300 into Cohort 1 (seat belt); 100 into Cohort 2 (distracted driving); 100 into Cohort 3 (drink driving). Each SMS intervention will be designed to target a single risk behavior. The study is powered to show a difference of 15% in the percentage of subjects reporting seat belt use at week 8. Other cohort trials (i.e. distracted driving, drink driving) and outcomes will be exploratory.

ELIGIBILITY:
Inclusion criteria:

1) Adult participant (age ≥ 18 years & ≤25 years)

1. Cohort 1: Any vehicle trip in past 2 weeks where individual reports not using a seat belt
2. Cohort 2: Any vehicle trip in past 2 weeks where individual reports phone was used to type while driving and car was moving
3. Cohort 3: Any vehicle trip in past 2 weeks where individual reports driving a vehicle within 2 hours after consuming 2 or more drinks

Exclusion criteria:

1. Member of a protected population (prisoner)
2. Unable to provide informed consent
3. No plan to drive and/or ride in a vehicle in the next month
4. Non-English speaking
5. No personal mobile phone or planning on changing phone in next 3 months

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pacella, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pennsylvania Hospital Emergency Departments, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Emergency Departments, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Procedures, including re-coding of key variables, will be put in place to allow for complete de-identification of the data. All relevant trial-related documents, including the protocol, data dictionary, and the main statistical code, will be shared along with the data. There will be no predetermined end date for the data sharing. Data will be available for any research purpose to all interested parties who have approval from an independent ethics review committee and who have a methodological sound proposal as determined by the steering committee of the current trial. Interested parties will be able to request the data by contacting the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after publication of main trial findings.
Access Criteria: Data will be available for any research purpose to all interested parties who have approval from an independent ethics review committee and who have a methodological sound proposal as determined by the steering committee of the current trial.

REFERENCES:
- [Derived] Suffoletto B, Pacella-LaBarbara ML, Huber J, Delgado MK, McDonald C. Effectiveness of a Text Message Intervention Promoting Seat Belt Use Among Young Adults: A Randomized Clinical Trial. JAMA Netw Open. 2022 Sep 1;5(9):e2231616. doi: 10.1001/jamanetworkopen.2022.31616. PMID 36129713

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SMS Intervention | SMS Assessments
Started | 110 | 108
Completed | 110 | 108
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMS Intervention | SMS Assessments | Total
Number analyzed (Participants) | 110 | 108 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.5 (2.2) | 21.6 (2.0) | 21.5 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 71 | 139
  Male | 42 | 37 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 37 | 35 | 72
  White | 51 | 60 | 111
  More than one race | 5 | 8 | 13
  Unknown or Not Reported | 10 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Seat Belt Use
Description: Participant count reporting always using a seat belt over past 2 weeks
Time Frame: Week 8
Population: 158 participants completed the 8-week follow-up and thus were included in outcome analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | SMS Intervention | SMS Assessments
Number analyzed (Participants) | 82 | 76
Participants | 34 | 15

2. Secondary Outcome: Feasibility of Recruitment
Description: Percentage of ED patients who screen positive
Time Frame: Baseline
Population: Reported less than always seat belt use in the past 2 weeks either as a driver or passenger and met other enrollment criteria
Measure: Count of Participants; unit: Participants
Groups:
- Screened Positive & Enrolled: Percentage of ED patients who screened positive for seat belt risk and met enrollment criteria
Arm/Group | Screened Positive & Enrolled
Number analyzed (Participants) | 702
Participants | 218

3. Secondary Outcome: Measure of Intervention Acceptability
Description: Percentage of ED patients enrolled in the Intervention arm who complete at least 50% of the SMS assessments during the intervention period
Time Frame: 2 weeks to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SMS Intervention | SMS Assessments
Number analyzed (Participants) | 110 | 108
Participants | 56 | 59

4. Secondary Outcome: Seat Belt Use
Description: Participant count reporting always using a seat belt over past 2 weeks
Time Frame: Week 14
Population: 140 participants completed the 14-week follow-up and thus were included in outcome analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | SMS Intervention | SMS Assessments
Number analyzed (Participants) | 75 | 65
Participants | 32 | 20

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | SMS Intervention | SMS Assessments
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/108
Other Adverse Events (participants affected / at risk) | 0/110 | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT03833713/Prot_SAP_001.pdf
  • Informed Consent Form (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT03833713/ICF_002.pdf